CLINICAL TRIAL: NCT05628428
Title: Effects of an Exercise Program on Cervical Pain Through Educational Videos: a Randomized Clinical Trial
Brief Title: Effects of Exercise on Cervical Pain Through Educational Videos
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Valencia (Other)
Responsible Party: Principal Investigator, David Hernández-Guillén, Assistant professor, PT, PhD, University of Valencia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: EX_ONLINE_01
Record Dates: First submitted 2022-11-15; First posted 2022-11-28 (Actual); Last update posted 2023-07-19 (Actual); Status verified 2023-07

CONDITIONS: Neck Pain
Keywords: Video pills; Exercise; Neck pain
MeSH Terms: conditions — Neck Pain; Motor Activity

STUDY DESIGN:
Intervention Model Description: Ramdomized clinical trial
Who Masked: Investigator, Outcomes Assessor
Masking Description: A researcher unrelated to the intervention will be responsible for randomizing the sample between the two groups. The researchers in charge of evaluating and interpreting the data will not know to which group each participant belongs.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise (Experimental): Exercising through educational videos for eight weeks. In addition, they will receive educational information about neck pain and the importance of exercise in this case, at the beginning of the study.
  Interventions: Other: Exercise to strengthen neck area.; Other: Information
- Control (Active Comparator): Educational information about neck pain and the importance of exercise in this case, at the beginning of the study.
  Interventions: Other: Information

INTERVENTIONS:
Other: Exercise to strengthen neck area. — An exercise protocol will be carried out through educational videos. There will be a total of four videos which will pose exercises for two weeks each. These exercises will be done twice a week. A reminder will be sent by email on the days that they must be carried out.
  Arms: Exercise
Other: Information — Information will be provided on neck pain and how exercise is able to help prevent it.

SUMMARY:
Due to the increased prevalence of neck pain in studied adolescents and young adults, this intervention is carried out, which mainly seeks to compare and verify the effectiveness of therapeutic exercise with education, compared to education alone.

It is also necessary to mention the high levels of stress levels reported in students, which can affect the increase in pain and the perception of these at times when stress increases. The intervention has been decreed in the weeks before and during the exam period at the University of Valencia, to see if the neck pain experienced by students at similar stages of their academic life is prevented or reduced.

It is decided to use education above all to give the participants a tool that allows the participants to find out what happens and why it happens when the participants suffer from neck pain, as well as an explanation of the pathology and the risk factors and how to avoid -the bear. In addition, knowledge about the condition in question can lead to a reconceptualization of pain, changing the approach and exposing a different approach, when treating the pathology.

It must be said that in the structure and layout of the informative document, the investigators think of an instrument that can serve the participants for the future.

Another reason for carrying out the study is the few tests on neck pain carried out with new technologies. The use of videos, therefore, seeks to facilitate access to the information provided, being a useful and practical tool for students, familiar with the use of new technologies.

In addition, the training is intended to be as didactic as possible, the chosen exercises are carefully explained and the fact that they are found in videos and not in a practical class, favors access to the content in these, for that the participants use the videos at their disposal. Finally, treating neck pain with training and education and taking into account the stress of students, brings to conventional treatment an interesting perspective of coping, focused on the biopsychosocial field.

ELIGIBILITY:
Inclusion Criteria:

* Students of first curse of physiotherapy.
* That they have had an episode of neck pain at exam time.

Exclusion Criteria:

* They do not want to sign the informed consent.
* That they present some pathology that causes chronic cervical pain.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2022-12-01 (Actual); Primary Completion 2023-04-30 (Actual); Study Completion 2023-05-31 (Actual)

PRIMARY OUTCOMES:
Visual Analogue Scale (VAS) | 0 week (baseline)
  Scale that evaluates pain from 0 to 10, where 0 means no pain and 10 means the worst pain imaginable.
Visual Analogue Scale (VAS) | 4 week (middle)
  Scale that evaluates pain from 0 to 10, where 0 means no pain and 10 means the worst pain imaginable.
Visual Analogue Scale (VAS) | 8 week (post intervention)
  Scale that evaluates pain from 0 to 10, where 0 means no pain and 10 means the worst pain imaginable.

SECONDARY OUTCOMES:
SISCO Inventory of Academic Stress | 0 week (baseline), 4 week, 8 week (post intervention)
  The SISCO Inventory is a measure of academic stress in students of upper education or postgraduates. Consists of 31 items including three broad factors: Stressors, Symptoms and Coping. The first item is intended to filter which respondents are suitable candidates to answer the questionnaire. The subsequent item measures the perceived intensity of academic stress. Stressors (first factor, 8 items) represent the frequency in which the demands of the environment are valued as stressors; Symptoms (second factor, 15 items) indicate the frequency in which the symptoms are presented; and Coping (third factor, 6 items), identify the frequency of coping strategies.
  Responses are provided on a 5-point Likert type scale anchored by 1 (never) to 5 (always).
Neck Disability Index | 0 week (baseline), 4 week, 8 week (post intervention)
  This questionnaire has been designed to give the doctor information as to how your neck pain has affected your ability to manage in everyday life. Questions are scored on a vertical scale of 0-5. Total scores and multiply by 2. Divide by number of sections answered multiplied by 10. A score of 22% or more is considered a significant activities of daily living disability.
EQ-5D-5L Quality of Life Questionnaire | 0 week (baseline), 4 week, 8 week (post intervention)
  This scale is divided into 5 items with 5 options each, which go from best to worst (1 best, 5 worst). In addition, a rule is used to assess health that goes from 0 to 100, where 0 is the worst possible health and 100 is the best possible health.

CONTACTS AND LOCATIONS:
Overall Officials: David Hernández-Guillén, PT, PhD, Principal Investigator — University of Valencia
Locations (1):
- Faculty of Physiotherapy of the University of Valencia, Valencia, Spain

IPD SHARING:
Plan to Share IPD: No